CLINICAL TRIAL: NCT03234881
Title: Weight Loss Treatment and CBT for Veterans With Binge Eating
Brief Title: Weight Loss Treatment for Veterans With Binge Eating
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIR 15-349
Record Dates: First submitted 2017-07-12; First posted 2017-07-31 (Actual); Results first posted 2024-06-28 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Binge Eating Disorder
Keywords: Binge Eating; Cognitive Behavioral Therapy; Weight Management; Veterans
MeSH Terms: conditions — Binge-Eating Disorder; Bulimia

STUDY DESIGN:
Intervention Model Description: This is a randomized RCT in which one half of participants will be assigned to MOVE! (treatment-as-usual weight management) and the other half will be assigned to MOVE! plus the experimental condition (clinician-led Cognitive Behavioral Therapy).
Who Masked: Care Provider
Masking Description: Treating therapists will be blind to outcome data
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MOVE! (Active Comparator): Weight management delivered as Treatment-as-Usual
  Interventions: Behavioral: MOVE!
- MOVE!+CBT (Experimental): Weight management delivered as Treatment-as-Usual plus use of a short duration, low-intensity CBT for recurrent binge eating.
  Interventions: Behavioral: MOVE!+CBT

INTERVENTIONS:
Behavioral: MOVE! — Participants randomized to the MOVE!(or TeleMOVE!) arm only. MOVE! is 16 weeks of 60-minute weekly groups that are led by a physical therapist, dietician, and/or clinical health psychologist. Clinicians utilize materials available online and encourage the use, but do not require or provide food diaries. TeleMOVE! is a 90-day program utilizing technology to provide home-based messaging focusing on health education and as needed clinician contact. *TeleMOVE! was added as an option since many in-person MOVE! programs were on pause due to the pandemic.
  Arms: MOVE!
Behavioral: MOVE!+CBT — Participants randomized to the MOVE!+CBT arm will attend the 16 weeks of 60-minute weekly MOVE! or 90-days of the TeleMOVE! Treatment groups, along with up to 10 clinician-led individual sessions over a 3-month period. Participants will also be given a patient treatment manual to read at home, food diaries that will be expected to be completed on a daily basis, and gradually increase daily physical activity.
  Arms: MOVE!+CBT

SUMMARY:
This study aims to adapt and test a cognitive behavioral therapy (CBT) treatment that can be administered concurrently with the Veteran's Health Administration (VHA) MOVE! weight management program for Veterans with DSM-5 Binge Eating Disorder (BED) and high weight.

DETAILED DESCRIPTION:
To date, there have been limited studies of Binge Eating Disorder (BED) and high weight utilizing combined eating disorder and weight management approaches in real-world settings, nor studies with complex and diverse samples. The objective of this project was to conduct a clinical trial that would produce evidence-based findings for a diverse patient group in a healthcare setting. Specifically, we aimed to address comorbid BED and high weight among Veterans in the Veteran's Health Administration (VHA), the largest integrated healthcare system in the U.S., by testing the effectiveness of VA's evidence-based weight management program, called MOVE!, versus MOVE! administered concurrent with a brief, clinician-led cognitive-behavioral therapy (CBT).

Aim 1: To assess the effectiveness of MOVE! (treatment-as-usual) to MOVE! plus brief, clinician-led CBT (MOVE!+CBT).

Hypothesis 1: It is hypothesized that MOVE!+CBT will have greater improvements on the primary outcomes of eating pathology and binge eating (reductions in binge frequency and percentage of participants who are binge remitted) than MOVE! alone.

Hypothesis 2: It is further hypothesized that MOVE!+CBT will have greater improvements on secondary measures of mental health, quality of life, and other eating behaviors.

Aim 2: To conduct exploratory analyses assessing the effectiveness of MOVE! to MOVE! vs. MOVE!+CBT on weight outcomes.

Hypothesis: It is hypothesized that MOVE!+CBT will have greater weight loss, and a larger percentage who achieve 5% weight loss, than MOVE! alone.

Note that several planned outcomes were not able to be analyzed for this project. Due to pandemic/COVID-19 related impacts, lipid profile data from in-person blood draws were inconsistently collected. Likewise, MOVE! adherence could not be measured with in-person session attendance as delivery for this intervention was expanded to include technology-delivered modalities. To fill these gaps, an "Impact of COVID-19" measure was added soon after the onset of the pandemic, but these questionnaire items did not hold up over the course of time and were removed. Finally, the 24-Hour Food Frequency Questionnaire (24 Hour-FFQ), a brief screening tool of food intake, was a measure specially designed for this study. Validation and publication of this screener was successful (The 24-hour food frequency assessment screening tool (FAST24): Development and evaluation of a novel dietary screener to identify foods associated with weight change - PubMed (nih.gov)), however, the lack of granular dietary data did not lend itself to measuring outcome. None of the measures removed represented primary or secondary outcomes for this project.

ELIGIBILITY:
Inclusion Criteria:

* BMI>=25
* Presence of recurrent binge eating on the MOVE! Survey

Exclusion Criteria:

* More than 4 MOVE! sessions in the prior year
* Active psychosis or suicidal ideation
* Medical or psychiatric illness, or cognitive deficits that interfere with providing consent or completing assessments
* Pregnancy or lactation

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2023-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robin M Masheb, PhD, Principal Investigator — VA Connecticut Healthcare System West Haven Campus, West Haven, CT
Locations (2):
- United States (2):
  - VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut
  - VA Central Western Massachusetts Healthcare System, Leeds, MA, Leeds, Massachusetts

IPD SHARING:
Plan to Share IPD: No
Unable to share Veteran data

REFERENCES:
- [Background] Masheb RM, Chan SH, Raffa SD, Ackermann R, Damschroder LJ, Estabrooks PA, Evans-Hudnall G, Evans NC, Histon T, Littman AJ, Moin T, Nelson KM, Pagoto S, Pronk NP, Tate DF, Goldstein MG. State of the art conference on weight management in VA: Policy and research recommendations for advancing behavioral interventions. J Gen Intern Med. 2017 Apr;32(Suppl 1):74-78. doi: 10.1007/s11606-016-3965-y. PMID 28271431
- [Result] Masheb RM, Douglas ME, Kutz AM, Marsh AG, Driscoll M. Pain and emotional eating: further investigation of the Yale Emotional Overeating Questionnaire in weight loss seeking patients. J Behav Med. 2020 Jun;43(3):479-486. doi: 10.1007/s10865-020-00143-4. Epub 2020 Feb 27. PMID 32107681
- [Result] Masheb RM, Snow JL, Fenn LM, Antoniadis NE, Raffa SD, Ruser CB, Buta E. Development and Psychometric Assessment of the Weight and Eating Quality of Life (WE-QOL) Scale in US Military Veterans. J Gen Intern Med. 2023 Jul;38(9):2076-2081. doi: 10.1007/s11606-023-08132-4. Epub 2023 Mar 27. PMID 36973571
- [Result] Carr MM, Lou R, Macdonald-Gagnon G, Peltier MR, Funaro MC, Martino S, Masheb RM. Weight change among patients engaged in medication treatment for opioid use disorder: a scoping review. Am J Drug Alcohol Abuse. 2023 Sep 3;49(5):551-565. doi: 10.1080/00952990.2023.2207720. Epub 2023 May 18. PMID 37200510
- [Result] Masheb RM, Buta E, Snow JL, Munro LF, Lawless M, Abel EA, McWain NE, Marsh A, Cary A, Grilo CM, Raffa SD, Ruser CB. Randomized Controlled Trial of Weight Management Versus Weight Management With Concurrent Cognitive-Behavioral Therapy for Binge-Eating Disorder in US Veterans With High Weight. Int J Eat Disord. 2025 Sep;58(9):1777-1792. doi: 10.1002/eat.24476. Epub 2025 Jun 9. PMID 40485646

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MOVE! | MOVE!+CBT
Started | 56 | 53
Completed | 47 | 50
Not Completed | 9 | 3
Not completed — Lost to Follow-up | 9 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MOVE! | MOVE!+CBT | Total
Number analyzed (Participants) | 56 | 53 | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (13.5) | 57.9 (10.5) | 55.8 (12.3)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex/Gender: Female | 11 | 16 | 27
  Sex/Gender: Male | 45 | 36 | 81
  Sex/Gender: Other, not specified | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 5 | 13
  Not Hispanic or Latino | 48 | 48 | 96
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Number analyzed is reflective of the number of participants that completed the assessment. Numbers differ from total number of participants since one participant chose not to answer this question.
  Participants
    Asian: number analyzed (Participants) | 55 | 53 | 108
    Asian | 0 | 1 | 1
    Black: number analyzed (Participants) | 55 | 53 | 108
    Black | 5 | 6 | 11
    More than one race/race not listed: number analyzed (Participants) | 55 | 53 | 108
    More than one race/race not listed | 3 | 2 | 5
    White: number analyzed (Participants) | 55 | 53 | 108
    White | 47 | 44 | 91
Education [Count of Participants; unit: Participants]
  >High School/High School | 7 | 12 | 19
  Some College | 27 | 16 | 43
  Completed College | 17 | 14 | 31
  Graduate School | 5 | 11 | 16
Married [Count of Participants; unit: Participants] | 28 | 29 | 57
Weight History [Mean (Standard Deviation); unit: lbs]
  Baseline Weight | 258 (50.2) | 249 (54.0) | 254 (52.0)
  Highest Adult Weight | 278 (52.9) | 266 (55.4) | 272 (54.2)
  Lowest Adult Weight | 170 (33.6) | 167 (37.1) | 168 (35.2)
Mental Health [Count of Participants; unit: Participants]
  Trauma (Positive PCL Criteria A) | 40 | 40 | 80
  Alcohol Use Disorder (Positive AUDIT-C) | 14 | 10 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change in Eating Disorder Examination-Self-report Questionnaire (EDE-Q)
Description: The EDE-Q is the self-report version of the more intensive EDE interview. Research has documented that the EDE-Q performs well as a measure of change in treatment trials and has adequate convergence with the interview format. The EDE-Q generates the same frequency data for eating behaviors (binge eating and overeating) in the past 28 days, and the same four subscales reflecting eating disorder pathology. Score on a scale 0-6; higher=worse
Time Frame: Pre treatment, 3 month post treatment, 9 month post treatment, 15 month post treatment
Population: Number analyzed for each timepoint is reflected below. Note some participants were lost to follow-up at each timepoint.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | MOVE! | MOVE!+CBT
Number analyzed (Participants) | 56 | 53
score on a scale
  Baseline | 3.18 (0.16) | 2.89 (0.19)
  3 Months: number analyzed (Participants) | 47 | 50
  3 Months | 2.81 (0.17) | 2.13 (0.17)
  9 Months: number analyzed (Participants) | 44 | 45
  9 Months | 2.57 (0.16) | 2.00 (0.19)
  15 Months: number analyzed (Participants) | 46 | 42
  15 Months | 2.50 (0.16) | 1.77 (0.19)

2. Primary Outcome: Change in Binge Episodes From Eating Disorder Examination Interview
Description: The EDE is a clinician administered interview that is considered to be the gold standard for diagnosing eating disorders and assessing binge frequency. Number of binges; higher=worse
Time Frame: Pre Treatment, 3 month post treatment, 9 month post treatment, 15 month post treatment
Population: Number analyzed for each timepoint is reflected below. Note some participants were lost to follow-up at each timepoint.
Measure: Mean (Standard Deviation); unit: Number of binges
Arm/Group | MOVE! | MOVE!+CBT
Number analyzed (Participants) | 56 | 53
Number of binges
  Baseline | 21.23 (19.03) | 21.75 (18.42)
  3 Months: number analyzed (Participants) | 46 | 50
  3 Months | 7.02 (8.62) | 3.64 (6.09)
  9 Months: number analyzed (Participants) | 43 | 45
  9 Months | 6.02 (7.3) | 5.38 (9.44)
  15 Months: number analyzed (Participants) | 41 | 41
  15 Months | 8.15 (10.77) | 6.98 (9.52)

3. Secondary Outcome: Change in Patient Health Questionnaire-9 (PHQ-9)
Description: The PHQ-9 is a 9-item version, is a self-report measure for the symptoms of depression. Score on scale from 0-27; higher=worse
Time Frame: Pre treatment, 3 month post treatment, 9 month post treatment, 15 month post treatment
Population: Number analyzed is reflective of the number of participants that completed the assessment at each timepoint. Numbers differ from each timepoint due to those that were lost to follow-up.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | MOVE! | MOVE!+CBT
Number analyzed (Participants) | 56 | 53
score on a scale
  Baseline | 9.44 (1.09) | 8.41 (0.94)
  3 Months: number analyzed (Participants) | 47 | 50
  3 Months | 7.89 (5.19) | 5.38 (0.73)
  9 Months: number analyzed (Participants) | 44 | 45
  9 Months | 7.95 (5.08) | 6.92 (1.00)
  15 Months: number analyzed (Participants) | 46 | 42
  15 Months | 7.47 (0.91) | 7.97 (5.04)

4. Secondary Outcome: Change in PTSD Checklist (PCL-5)
Description: The PCL-5 is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of Post Traumatic Stress Disorder (PTSD). Score on scale from 0-80; higher=worse
Time Frame: Pre treatment, 3 month post treatment, 9 month post treatment, 15 month post treatment
Population: as for outcome 3
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | MOVE! | MOVE!+CBT
Number analyzed (Participants) | 56 | 53
score on a scale
  Baseline | 37.48 (3.76) | 31.27 (4.11)
  3 Months: number analyzed (Participants) | 47 | 50
  3 Months | 27.67 (2.85) | 22.62 (3.00)
  9 Months: number analyzed (Participants) | 44 | 45
  9 Months | 29.29 (3.36) | 28.46 (3.60)
  15 Months: number analyzed (Participants) | 46 | 42
  15 Months | 27.05 (3.57) | 23.85 (3.67)

5. Secondary Outcome: Weight and Eating Quality of Life (WE-QoL)
Description: The WE-QoL is an 8-item self-report instrument for measurement of the impact weight and eating has on quality-of-life outcomes. Score on scale from 0-4; higher=worse
Time Frame: Pre Treatment, 3 month post treatment, 9 month post treatment, 15 month post treatment
Population: as for outcome 3
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | MOVE! | MOVE!+CBT
Number analyzed (Participants) | 56 | 53
score on a scale
  Baseline | 1.58 (0.12) | 1.50 (0.14)
  3 Months: number analyzed (Participants) | 47 | 50
  3 Months | 1.29 (0.16) | 1.12 (0.14)
  9 Months: number analyzed (Participants) | 44 | 45
  9 Months | 1.33 (0.16) | 1.05 (0.16)
  15 Months: number analyzed (Participants) | 46 | 42
  15 Months | 1.18 (0.17) | 1.01 (0.14)

6. Secondary Outcome: Change in European Quality of Life (EuroQoL-5D)
Description: The EuroQol-5D is a 5-item self-report instrument for measurement of quality of life outcomes that has specifically been used in weight loss trials with Veterans. The EuroQoL-5D also includes the Visual Analogue Scale (VAS) which is a measure of overall self-rated health status on a 100-point scale. Units on a scale (0-100); higher=better
Time Frame: Pre treatment, 3 month post treatment, 9 month post treatment, 15 month post treatment
Population: as for outcome 3
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | MOVE! | MOVE!+CBT
Number analyzed (Participants) | 56 | 53
units on a scale
  Baseline | 56.8 (2.64) | 52.8 (2.94)
  3 Months: number analyzed (Participants) | 47 | 50
  3 Months | 63 (2.73) | 69.05 (2.57)
  9 Months: number analyzed (Participants) | 44 | 45
  9 Months | 66.35 (2.88) | 68.07 (2.72)
  15 Months: number analyzed (Participants) | 46 | 42
  15 Months | 66.27 (3.29) | 63.54 (3.22)

7. Secondary Outcome: Night Eating Questionnaire (NEQ)
Description: The NEQ is a 14-item self-report instrument for the measurement of Night Eating Syndrome (NES). A total score of greater than or equal to 25 indicates NES. Score on scale 0-52; higher=worse
Time Frame: Pre Treatment, 3 month post treatment, 9 month post treatment, 15 month post treatment
Population: as for outcome 3
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | MOVE! | MOVE!+CBT
Number analyzed (Participants) | 56 | 53
score on a scale
  Baseline | 21.06 (1.24) | 21.25 (1.37)
  3 Months: number analyzed (Participants) | 47 | 50
  3 Months | 18.89 (1.29) | 15.70 (1.27)
  9 Months: number analyzed (Participants) | 44 | 45
  9 Months | 17.89 (1.18) | 16.98 (1.27)
  15 Months: number analyzed (Participants) | 46 | 42
  15 Months | 18.06 (1.20) | 16.90 (1.07)

8. Secondary Outcome: CBT Session Attendance (Treatment Dose)
Description: CBT session attendance will be determined by the number of clinician-led individual sessions attended throughout the treatment.
Time Frame: 3 month post-treatment
Measure: Mean (Full Range); unit: number of sessions
Arm/Group | MOVE!+CBT
Number analyzed (Participants) | 50
number of sessions | 7.75 [0 to 9]

9. Other Pre Specified Outcome: Change in BMI
Description: BMI will be calculated based upon self-reported height and weight. A BMI of 25.0-29.9 indicates overweight, and 30.0 above indicates obesity. Kg/m 2; higher=worse
Time Frame: Pre treatment, 3 month post treatment, 9 month post treatment, 15 month post treatment
Population: as for outcome 3
Measure: Mean (Standard Error); unit: kg/m^2
Arm/Group | MOVE! | MOVE!+CBT
Number analyzed (Participants) | 56 | 53
kg/m^2
  Baseline | 38.17 (1.20) | 35.58 (0.94)
  3 Months: number analyzed (Participants) | 47 | 50
  3 Months | 37.24 (1.24) | 34.52 (0.96)
  6 Months: number analyzed (Participants) | 44 | 45
  6 Months | 36.58 (1.28) | 34.21 (0.91)
  9 Months: number analyzed (Participants) | 46 | 42
  9 Months | 36.55 (1.25) | 34.23 (0.89)

10. Other Pre Specified Outcome: Change in Weight Control Strategies Scale (WCSS)
Description: The WCSS is a self-report instrument that assesses the use of specific weight loss behaviors. The measure has been shown to be valid, reliable and predictive of weight loss. Score on a scale 0-4; higher=better
Time Frame: Pre treatment, 3 month post treatment, 9 month post treatment, 15 month post treatment
Population: as for outcome 3
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | MOVE! | MOVE!+CBT
Number analyzed (Participants) | 56 | 53
score on a scale
  Baseline | 1.49 (0.08) | 1.62 (0.09)
  3 Months: number analyzed (Participants) | 47 | 50
  3 Months | 1.81 (0.1) | 2.18 (0.1)
  9 Months: number analyzed (Participants) | 44 | 45
  9 Months | 1.77 (0.1) | 1.83 (0.1)
  15 Months: number analyzed (Participants) | 46 | 42
  15 Months | 1.8 (0.1) | 1.71 (0.1)

11. Other Pre Specified Outcome: Change in Godin Leisure Time Exercise Questionnaire (Godin)
Description: The Godin is a 4-item, reliable self-report measure of physical activity that assesses the frequencies of strenuous, moderate and mild exercise and has been validated against accelerometers. Units on a scale 0-119; higher=better
Time Frame: Pre treatment, 3 month post treatment, 9 month post treatment, 15 month post treatment
Population: as for outcome 3
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | MOVE! | MOVE!+CBT
Number analyzed (Participants) | 56 | 53
score on a scale
  Baseline | 21.36 (3.45) | 26.93 (3.82)
  3 Months: number analyzed (Participants) | 47 | 50
  3 Months | 27.91 (4.43) | 32.49 (3.51)
  9 Months: number analyzed (Participants) | 44 | 45
  9 Months | 30 (3.68) | 25.19 (4.20)
  15 Months: number analyzed (Participants) | 46 | 42
  15 Months | 28.46 (3.75) | 25.95 (3.78)

12. Other Pre Specified Outcome: Treatment Satisfaction
Description: Treatment satisfaction will be measured with a number of questions to measure participants' experience as a participant on a range from strongly disagree to strongly agree (e.g., "I increased my ability to manage my binge eating" and "How likely are you to recommend this treatment to other Veterans?"). Score on a scale 0-48; higher=better
Time Frame: 3 months post treatment
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | MOVE! | MOVE!+CBT
Number analyzed (Participants) | 47 | 50
score on a scale | 34.43 (1.39) | 40.94 (0.77)

13. Other Pre Specified Outcome: Change in Weight
Description: All weights were taken by self-report at each timepoint.
Time Frame: Pre Treatment, 3 month post treatment, 9 month post treatment, 15 month post treatment
Population: as for outcome 3
Measure: Mean (Standard Error); unit: lbs
Arm/Group | MOVE! | MOVE!+CBT
Number analyzed (Participants) | 56 | 53
lbs
  Baseline | 253.83 (9.32) | 235.11 (7.41)
  3 Months: number analyzed (Participants) | 47 | 50
  3 Months | 247.67 (9.43) | 227.87 (7.12)
  9 Months: number analyzed (Participants) | 44 | 45
  9 Months | 243.59 (9.96) | 225.94 (7.06)
  15 Months: number analyzed (Participants) | 46 | 42
  15 Months | 243.24 (9.67) | 226.33 (7.11)

14. Other Pre Specified Outcome: Loss of Control Overeating Scale (LOCES)
Description: A self-administered scale used to assess features of loss of control over eating. Score on a scale 0-4; higher=worse
Time Frame: Pre Treatment, 3 month post treatment, 9 month post treatment, 15 month post treatment
Population: as for outcome 3
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | MOVE! | MOVE!+CBT
Number analyzed (Participants) | 56 | 53
score on a scale
  Baseline | 2.64 (0.18) | 2.21 (0.18)
  3 Months: number analyzed (Participants) | 47 | 50
  3 Months | 1.70 (0.20) | 1.14 (0.17)
  9 Months: number analyzed (Participants) | 44 | 45
  9 Months | 1.62 (0.17) | 1.11 (0.17)
  15 Months: number analyzed (Participants) | 46 | 42
  15 Months | 1.58 (0.21) | 1.17 (0.19)

15. Other Pre Specified Outcome: Modified Yale Food Addiction Scale 2.0 (mYFAS 2.0)
Description: A self-administered scale used to assess the features of food addiction. Units on a scale 0-11; higher=worse
Time Frame: Pre Treatment, 3 month post treatment, 9 month post treatment, 15 month post treatment
Population: as for outcome 3
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | MOVE! | MOVE!+CBT
Number analyzed (Participants) | 56 | 53
units on a scale
  Baseline | 4.73 (0.46) | 4.28 (0.52)
  3 Months: number analyzed (Participants) | 47 | 50
  3 Months | 3.02 (0.37) | 2.35 (0.35)
  9 Months: number analyzed (Participants) | 44 | 45
  9 Months | 2.75 (0.47) | 2.96 (0.46)
  15 Months: number analyzed (Participants) | 46 | 42
  15 Months | 2.53 (0.45) | 2.49 (0.44)

ADVERSE EVENTS:
Time Frame: AEs, SAEs, and UAPs were collected from the time of study entry until the end of study participation (a total of 15 months)
Description: The overall risk for this study was minimal. The risks associated with assessments are only minor due to an inconvenience that may occur during their completion (frustrating/time-consuming). Risks associated with treatments may include no benefit or worsening of binge eating.
Arm/Group | MOVE! | MOVE!+CBT
All-Cause Mortality (participants affected / at risk) | 1/56 | 0/53
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/53
Other Adverse Events (participants affected / at risk) | 0/56 | 0/53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-16): https://cdn.clinicaltrials.gov/large-docs/81/NCT03234881/Prot_SAP_000.pdf